CLINICAL TRIAL: NCT06986538
Title: A Multicenter Randomized Controlled Study of the Extent of Lymph Node Dissection for Advanced Right-sided Colon Cancer
Brief Title: Extent of Lymph Node Dissection for Advanced Right-Sided Colon Cance
Acronym: MARCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MARCH
Record Dates: First submitted 2025-04-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Advanced Right-sided Colon Cancer; the Extent of Lymph Node Dissection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMV group (Active Comparator)
  Interventions: Procedure: Clearance with the left side of the SMV as the medial boundary
- SMA group (Experimental)
  Interventions: Procedure: Clearance with the left side of the SMA as the medial boundary

INTERVENTIONS:
Procedure: Clearance with the left side of the SMV as the medial boundary — Undergo radical resection for right colon cancer with the left side of the SMV as the medial boundary
  Arms: SMV group
Procedure: Clearance with the left side of the SMA as the medial boundary — Undergo radical resection for right colon cancer with the left side of the SMA as the medial boundary
  Arms: SMA group

SUMMARY:
This is a prospective multicenter randomized controlled clinical study to explore the extent of lymph node dissection in progressive right hemicolon cancer and to elucidate the pattern of lymphatic drainage in the right hemicolon.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years
2. Preoperative pathologic confirmation of adenocarcinoma
3. Tumor located in the region from the ileocecal valve to the right one-third of the transverse colon
4. American Society of Anesthesiologists (ASA) physical status classification I to III
5. Patients who have not received preoperative radiotherapy, chemotherapy, or immunotherapy
6. Preoperative imaging staging cT4N0M0 or cT3-4N+M0
7. Willing to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Past medical history of malignant tumor
2. Patients with multiple primary tumors
3. Patients with a history of inflammatory bowel disease or familial adenomatous polyposis
4. Patients with distant metastasis
5. Pregnant or breastfeeding women
6. History of other previous major abdominal surgery
7. Patients requiring emergency surgery (including tumor perforation, obstruction, hemorrhage, etc.)
8. Those with other clinical and laboratory conditions deemed by the investigator to be inappropriate for participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1064 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | The third postoperative year
  It is defined as the proportion of patients from the start of randomization to the end of the third year without any of the following events: disease progression, local recurrence, distant metastasis, second primary colorectal cancer, or death from any cause.

SECONDARY OUTCOMES:
overall survival | The third postoperative year
  The time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Cancer Hospital, Chinese Academyof Medical Sciences, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Affiliated Union Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Department of Coloretcal Surgery, the Sixth Affiliated Hospital of Sun Yat-sen University,, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Zhaoqing First People's Hospital, Zhaoqing, Guangdong
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospita, Shanghai, Shanghai Municipality
  - Changhai Hospitalof Naval Medical University, Shanghai, Shanghai Municipality
  - Shaanxi ProvincialPeople's Hospital, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of WenzhouMedical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No